CLINICAL TRIAL: NCT01328860
Title: Safety of Autologous Stem Cell Treatment for Spinal Cord Injury in Children
Brief Title: Autologous Stem Cells for Spinal Cord Injury (SCI) in Children
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator relocated to Orlando, Florida.
Sponsor: Aryn Knight (Other)
Collaborators: The Institute for Rehabilitaion and Research Foundation (Other); The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center (Other); Baylor College of Medicine (Other); Florida Hospital for Children (Other)
Responsible Party: Sponsor-Investigator, Aryn Knight, AVP Research, Memorial Hermann Health System
Organization: Memorial Hermann Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBIND14281
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injury
Keywords: Autologous; Stem Cells; Spinal Cord Injury; Children
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biologic; Stem Cells (Experimental)
  Interventions: Biological: bone marrow progenitor cells (BMPC) autologous transplantation

INTERVENTIONS:
Biological: bone marrow progenitor cells (BMPC) autologous transplantation — Not more than 5ml/kg bone marrow will be collected under anesthesia; after the bone marrow has been processed, about 6-8 hours after bone marrow aspiration, subjects will receive the cells via intra-venous (in the vein) infusion and will be monitored for 24 hours for any adverse events.
  Other Names: Autologous Stem Cells; Patient's own Stem Cells

SUMMARY:
The purpose of this research study is:

1. To see if Bone Marrow Cell harvest and transplantation are safe in children with Spinal Cord Injury, and
2. To determine if late functional outcome is improved following Bone Marrow Cell transplantation in children with Spinal Cord Injury, using pre-transplantation spinal cord function as the control.

DETAILED DESCRIPTION:
Of the estimated 11,000 cases of acute spinal cord injury (SCI) which occur each year in North America, 5% involve children. The injury is divided into the primary mechanical event which causes the injury, and the secondary events which follow. Outcome for SCI depends of the severity of the primary injury (complete vs. incomplete) and the spinal cord level of the injury. Current therapy is designed only to minimize the secondary events of SCI and other trauma-associated injuries. Because the current therapy does nothing to reverse the primary insult, significant advances in reducing the disability associated with SCI are unlikely. Recent basic science and animal studies suggest that stem cell treatment can foster functional improvement after SCI by helping repair the primary injury and reducing the secondary injury.

Stem cells are "unspecialized" cells in the body that do not have a specific function yet (for example, they have not become "heart cells" or "brain cells" yet.) Stem cells are able to divide and develop into more mature, function-specific cells and take the place of those cells that die, are injured or can no longer function the way they are supposed to. Stem cells are being studied a lot because of this ability and there is the possibility that they may be used to take the place of cells that are no longer working in different parts of the body because of disease (as in cancer, diabetes, and heart disease). Stem cells can be found throughout the body, but they are most common in the bone marrow, the thick, spongy material inside the bones.

The primary objective of this study is to determine the safety of transplantation of the patient's own (autologous) Bone Marrow Progenitor Cells (BMPC) in children with SCI. The secondary objective is to determine if functional, physiological and anatomic outcome measures are improved after BMPC autologous transplantation in children with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Between 1 year and 15 years of age on the day of study BMPC infusion.
2. Survived at least six months with PSCI, but are less than 4 years post injury (± 30 days), and have fixed neurologic deficits related to their injury at the time of enrollment.
3. Ability of child to understand and speak English.
4. Ability of child and caregiver to travel to Houston, Texas, and stay for at least 4 days, and to return for all Follow-up visits (patient is responsible for cost of travel and lodging while in Houston).
5. Pediatric patients with any type of spinal cord injury as long as their spinal cords are continuous on MRI evaluation. This includes paraplegic and quadriplegic patients with complete or incomplete spinal cord injuries. This includes patients with ASIA impairment scales from A to D. The clinical classification will be described by the level below which motor/sensory function is impaired, and the degree of that impairment. (i.e. C-5 if the deltoid muscle is intact but the biceps and other muscle groups below the C-5 level are weak [incomplete motor injury] or paralyzed [complete motor injury]. A similar evaluation of sensory function will be established clinically.

Exclusion Criteria:

1. Lack of informed consent.
2. Uncorrected coagulopathy during the baseline period defined as: INR > 1.4; PTT > 35 sec; PLT < 100,000.
3. Pre-injury history of seizure disorder and/or neurological impairment where the patient would not be able to participate in age appropriate pain rating scales.
4. A history of prior SCI or severe traumatic brain injury.
5. Known history of:

   * Recently diagnosed infection (within past 2 weeks) requiring treatment and/or medical intervention.
   * Renal disease or altered renal function as defined by serum creatinine > 1.5 mg/dL.
   * Hepatic disease or altered liver function as defined by SGPT > 150 U/L, and/or T. Bilirubin > 1.3 mg/dL.
   * Malignancy.
   * Immunosuppression as defined by WBC < 3 (10x3) at screening and/or baseline evaluation lab.
   * HIV.
   * Hepatitis B or C.

8. Unhealed fractures or wounds including osteomyelitis.

9. Pneumonia, or chronic lung disease requiring oxygen.

10. An anatomically discontinuous spinal cord diagnosed by CT or MRI imaging.

11. Positive urine pregnancy test (urine pregnancy test will be routinely performed on females of childbearing potential, age 11 or older.

12. Participation in a concurrent intervention study.

13. Desire for organ-donation in the event of death.

14. Unwillingness or inability to stay for at least four days following BMPC infusion (should any problems arise following the infusion) and to return for a 30 day, and 6 month follow-up visit, and be available for 1 year, and 2 year follow-up phone calls.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) - Standard Neurological Classification of Spinal Cord Injury. | 180 days
  ASIA classification assessment will take place pre-procedure, 1 day, 30 days, and 180 days post-procedure to define changes in functional outcome.

SECONDARY OUTCOMES:
Standard Neuropathic Pain Rating Scale | 2 years
  Assessment for improvement, worsening or development of neuropathic pain with an age appropriate standard pain rating scale will be performed pre-procedure, and post-procedure days 1 - 14, and again 30 days, 180 days, 1 year, and 2 year post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: James E. Baumgartner, MD, Study Chair — MHHS, Houston,TX & FL Hospital for Children, Orlando, FL; Rex A. Marco, MD, Principal Investigator — University of Texas Health Science Center, Houston TX
Locations (1):
- Children's Memorial Hemann Hospital; University of Texas Health Science Center - Houston, Houston, Texas, United States